CLINICAL TRIAL: NCT03534193
Title: Effectiveness of Using Educational Modules Via Bedside Tablet in Newly Diagnosed Type 1 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Site resources
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Verizon Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO 2016-0713
Record Dates: First submitted 2018-05-09; First posted 2018-05-23 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of 2 arms:
  Group 1 - standard Diabetic education-consisting of one on one education with a Registered Nurse in addition to the Molly Center Diabetes Care Guide (paper based) Group 2 - standard Diabetic education plus Bedside tablet with interactive Diabetic modules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Diabetic Education (Other): Participants randomized to Group 1 will receive Standard Diabetic Education with Registered Nurse and Molly Center Diabetes Care Guide (paper-based)
  Interventions: Other: Molly Center Diabetes Care Guide (Paper-based)
- Standard Diabetes Education and Tablet (Experimental): Participants randomized to Group 2 will receive Molly Center Standard Diabetes Education plus access to Tablet based interactive diabetes education modules
  Interventions: Other: Molly Center Diabetes Care Guide (Paper-based); Other: Tablet based interactive diabetes education modules

INTERVENTIONS:
Other: Molly Center Diabetes Care Guide (Paper-based) — Diabetes education with Registered Nurse in addition to Paper based education modules
Other: Tablet based interactive diabetes education modules — Molly Center Standard Diabetes Education plus access to interactive diabetes education modules through bedside tablet.
  Arms: Standard Diabetes Education and Tablet

SUMMARY:
This is a prospective, randomized trial to evaluate the effectiveness of using educational modules accessed through a bedside tablet in patients newly diagnosed with Type 1 Diabetes as an adjunct to *standard Children's Hospital- Molly Center diabetes education in comparison to *standard Children's Hospital- Molly Center diabetes education. (standard diabetes education consists of paper based reading material and nursing education).

DETAILED DESCRIPTION:
Type I diabetes is one of the most common diseases of childhood and its incidence has been increasing worldwide. By age 18, 1 in 300 children will be affected by Type 1 Diabetes1. Not only are children diagnosed with diabetes met with significant morbidity due to their disease, but they are also expected to be active participants in daily often complicated treatment regimens. As children with Type 1 diabetes grow older and eventually spend time away from their parents or caregivers, they are forced to manage their own care. Over the last several years, health systems in the United States have become more patient-centered and have focused on autonomy and patient preference. With the advent of technology that makes self-directed education possible, this patient-centered approach needs to be applied to children diagnosed with Type I diabetes.

When clinicians are at the center of educating patients with diabetes, they often communicate more directly with parents, who then use the information they receive to manage their child's care. This model, however, does not account for the fact that children with diabetes will one day need to manage their own care and that patients who are active participants and who understand their disease process will be more likely to cooperate with treatment regimens and lifestyle interventions. It is often difficult for any patient, child or adult, to process educational information provided verbally in a physician's office, especially immediately after they have been diagnosed with a life-long disease. Educational tools therefore need to focus on incorporating methods that best serve the patients being educated.

Since individuals learn in different ways and at different paces, interactive educational tools can help patients and their families learn in a way that can be individualized and private and can also be fun and creative. As our patients are growing up surrounded by technology, the use of this technology for education might provide a sense of normalcy to children and teenagers already overwhelmed by processes that are often difficult for them to identify with or understand. We hope that patients and families who are given the opportunity to learn independently will become better equipped to manage self-care and will develop a sense of involvement in their treatment. Interactive tools will also help patients and families become more actively engaged in understanding their disease process and can help them to become more active participants in their care.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosed Type 1 Diabetes admitted to the Joseph M. Sanzari Children's Hospital
* Patient/Caretaker/Family willing to complete questionnaires

Exclusion Criteria:

* Patients with previous history of Diabetes
* Patients with no plans to follow up at The Joseph M. Sanzari Children's Hospital - Molly's Center for Children with Diabetes and Endocrine Disorders after hospital discharge
* Non English speaking patients/family/caretaker

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2025-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Ghanny, MD, Principal Investigator — Joseph M.Sanzari Children's Hospital at Hackensack University Medical Center
Locations (1):
- Joseph M. Sanzari Children's Hospital, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Diabetes Education: Participants randomized to Group 1 will receive Standard Diabetic Education with Registered Nurse and Molly Center Diabetes Care Guide (paper-based)
  Molly Center Diabetes Care Guide (Paper-based): Diabetes education with Registered Nurse in addition to Paper based education modules
Period: Overall Study
Arm/Group | Standard Diabetes Education | Standard Diabetes Education and Tablet
Started | 14 | 14
Completed | 13 | 11
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Diabetes Education | Standard Diabetes Education and Tablet | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 14 | 28
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 9.78 [3 to 17] | 8.85 [2 to 17] | 9.31 [2 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 5 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 7 | 9 | 16
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 11 | 19
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Tablet Education in Newly Diagnosed Type 1 Diabetes
Description: Effectiveness of tablet education modules as measured by a diabetic knowledge post-test questionnaire.
  Total score ranges from 0-100%, with a higher percentage on the scale indicating a better outcome/knowledge.
Time Frame: Test will be completed on day 3 (+/- 2 days)
Population: post-education test score (percentile of questions answered correctly)
Measure: Mean (Full Range); unit: percentage of questions answered correct
Arm/Group | Standard Diabetes Education | Standard Diabetes Education and Tablet
Number analyzed (Participants) | 13 | 11
percentage of questions answered correct | 83 [70 to 90] | 86 [70 to 90]

2. Secondary Outcome: Improved Subject Compliance With Glucose Monitoring A1 Levels
Description: Subjects randomized to tablet education modules will demonstrate improved compliance with glucose monitoring as measured by Lower Hemoglobin A1C at initial follow up visit
Time Frame: Assessements will occur at 3 months
Population: lower HbA1C comparing to baseline
Measure: Mean (Full Range); unit: percentage change in HbA1C
Arm/Group | Standard Diabetes Education | Standard Diabetes Education and Tablet
Number analyzed (Participants) | 13 | 11
percentage change in HbA1C | 8 [7.1 to 14] | 8.06 [5.9 to 10.1]

3. Secondary Outcome: Improved Subject Compliance With Glucose Monitoring - Hypoglycemic Episodes
Description: Subjects randomized to tablet education modules will demonstrate improved compliance with glucose monitoring as measured by lower number of hypoglycemic episodes before initial follow up visit
Time Frame: Assessements will occur at 3 months
Population: number of Hypoglycemic Episodes
Measure: Mean (Full Range); unit: number of Hypoglycemic Episodes
Arm/Group | Standard Diabetes Education | Standard Diabetes Education and Tablet
Number analyzed (Participants) | 13 | 11
number of Hypoglycemic Episodes | 4.2 [0 to 15] | 1 [0 to 5]

4. Secondary Outcome: Improved Subject Compliance With Glucose Monitoring - Compliance With Daily Blood Glucose Monitoring
Description: Subjects randomized to tablet education modules will demonstrate improved compliance with glucose monitoring as measured by compliance with daily blood glucose monitoring at initial follow up visit
Time Frame: Assessements will occur at 3 months
Population: Number of times blood sugar was checked. Data was not collected as patients did not report it for either group.
Arm/Group | Standard Diabetes Education | Standard Diabetes Education and Tablet
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up until study completion (3 months +/- 20 days)
Arm/Group | Standard Diabetes Education | Standard Diabetes Education and Tablet
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11

LIMITATIONS AND CAVEATS:
The team experienced difficulties in collecting the number of blood sugar checks from the patients who did not report it for either group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/93/NCT03534193/Prot_000.pdf